CLINICAL TRIAL: NCT05876494
Title: Serum Lactate and Mean Platelet Volume as Predicators for Acute Exacerbation in Patients With Ulcerative Colitis
Brief Title: Serum Lactate and Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abu Elfatth, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: Alaa Esam
Record Dates: First submitted 2023-05-07; First posted 2023-05-25 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with ulcerative colitis: any patients with ulcerative colitis
  Interventions: Diagnostic Test: serum lactate

INTERVENTIONS:
Diagnostic Test: serum lactate — assessment of serum lactate and mean platelets volume

SUMMARY:
Patients presenting with severe symptoms of ulcerative colitis (UC) require hospital admission for urgent assessment and therapy. Endoscopic examination of the rectum and/or distal colon is often performed to assess severity and obtain tissue for histopathologic evaluation, but this is often extended to full colonoscopy to assess the extent of bowel involvement. Full colonoscopy is hazardous in this setting

DETAILED DESCRIPTION:
Biomarkers like erythrocyte sedimentation rate (ESR) and C reactive protein (CRP) are used for monitoring the disease activity but present a low specificity and sensitivity in UC . There are fecal biomarkers with better performance for detecting disease activity in UC like fecal calprotectin and lactoferrin, however, are very expensive Platelets present granules with Interleukin 8 (IL-8) which is a potent neutrophil chemoattractant and its cytoplasm contains P-selectin that induces overproduction of superoxide and the formation of neutrophil-platelet aggregates, which are elevated in patients with UC. The inhibition of this aggregates suppress the appearance of colon inflammation

The mean platelet volume (MPV) is correlated to the UC activity as also the increase of white blood count (WBC) mainly neutrophils. The interaction of neutrophil-platelet is a possible explanation of the high prevalence of thrombosis in UC due to the formation of Neutrophil Extracellular Traps (NETs) through Toll-like receptor 4 (TLR-4)

ELIGIBILITY:
Inclusion criteria:

Any patient who is above age of 18 years old and diagnosed to have UC based on combination between clinical, laboratory, radiological, endoscopic and/or histopathological data whatever the course of the disease Exclusion criteria

* Patients with inflammatory bowel disease (IBD) other than UC as those with Crohn's disease or microscopic colitis
* Pregnant patients with ulcerative colitis.
* Patients with UC who are under age of 18 years old
* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who is above age of 18 years old and diagnosed to have UC based on combination between clinical, laboratory, radiological, endoscopic and/or histopathological data whatever the course of the disease
Sampling Method: Non-Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy (%) of serum lactate in prediction the acute flare of ulcerative colitis | one year
  By using the receiver operator characteristics curve, we can determine the best cutoff point of serum lactate to predict the acute flare of ulcerative colitis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abu-Elfatth, Principal Investigator — Assiut University
Locations (1):
- Ahmed Mohammed Abu-Elfatth, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not yet

REFERENCES:
- [Background] Bennike T, Birkelund S, Stensballe A, Andersen V. Biomarkers in inflammatory bowel diseases: current status and proteomics identification strategies. World J Gastroenterol. 2014 Mar 28;20(12):3231-44. doi: 10.3748/wjg.v20.i12.3231. PMID 24696607